CLINICAL TRIAL: NCT00920413
Title: Randomized, Double-Blind, Placebo-Controlled Trial of Oral Vitamin C on Correction of Anemia in Patients Receiving Peritoneal Dialysis
Brief Title: Oral Vitamin C for Correction of Anemia in Patients Receiving Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Dr. Lori MacCallum, St. Michael's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-044
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2009-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Anemia; Peritoneal Dialysis
MeSH Terms: conditions — Anemia | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin C (Active Comparator): vitamin C 500mg orally once a day
  Interventions: Dietary Supplement: Vitamin C
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — vitamin C 500mg orally once a day
  Arms: vitamin C
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
People with kidney failure are at risk for the development of anemia. Anemia is a decrease in the production of hemoglobin, a substance that carries oxygen in the blood. The majority of patients require erythropoietin and iron supplementation to correct the anemia. In some patients, the hemoglobin fails to rise to a desired level despite treatment with erythropoietin and iron. There have been several studies in hemodialysis patients showing that vitamin C given intravenously helps to correct anemia in patients already on erythropoietin and iron.

The purpose of this study is to determine whether oral vitamin C will improve parameters of anemia in patients receiving peritoneal dialysis.

Description of the research

This is a randomized, double blind, placebo controlled study. Participants will be randomized in a 1:1 ratio to oral vitamin C 500mg once a day or placebo for 3 months. All participants will be receiving oral iron supplementation, subcutaneous erythropoietin and a B and C complex vitamin containing 100mg of vitamin C. Lab parameters (hemoglobin, TSAT, ferritin) will be done at baseline and then monthly. The primary outcome is percent change from baseline in transferrin saturation. Secondary objectives are percent change in ferritin, hemoglobin and erythropoietin dose from baseline.

DETAILED DESCRIPTION:
Patients will be randomized in a 1:1 ratio to Vitamin C 500mg orally once daily or matching placebo for 3 months. Randomization codes will be kept by the Research Pharmacy and investigators and patients will be blinded to treatment. Patients currently taking vitamin C supplements (excluding the 100mg of vitamin C contained in a B and C complex vitamin, a supplement used by all peritoneal dialysis patients), will be taken off the vitamin C and then randomized to one of the treatment arms after a 1 month washout period. At the end of 3 months, the effects of vitamin C on the change in transferrin saturation from baseline will be evaluated to identify which patients, if any, benefited from treatment. Hemoglobin, serum iron, total iron binding capacity, ferritin, transferrin saturation and erythropoietin dose will also be assessed. The dose and formulation of recombinant erythropoietin and oral iron will be adjusted during the study period according to standard practice algorithms currently used in the clinic. The addition of vitamin C does not pose any risk to the patients and will be dispensed to the patient by the Research Pharmacy at St. Michael's Hospital free of charge.

Patient population Inclusion criteria Receiving peritoneal dialysis for 2 months

Exclusion criteria Red blood cell folate < 3.9 nmol/L Serum B12 <110 pmol/L Bleeding, blood transfusions, acute liver disease in the previous 3 months

Assessments Parathyroid hormone Baseline B12 Baseline Folate Baseline Hemoglobin Baseline and monthly Hematocrit Baseline and monthly Ferritin Baseline and monthly Transferrin saturation Baseline and monthly Serum iron Baseline and monthly

ELIGIBILITY:
Inclusion Criteria:

* Receiving peritoneal dialysis for 2 months

Exclusion Criteria:

Red blood cell folate < 3.9 nmol/L

* Serum B12 <110 pmol/L
* Bleeding, blood transfusions, acute liver disease in the previous 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-03

PRIMARY OUTCOMES:
difference in percent change from baseline to 3 months in transferrin saturation between vitamin C and placebo | 3 months

SECONDARY OUTCOMES:
difference in percent change from baseline to 3 months in hemoglobin,ferritin and epoetin dose (each determined separately) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori A MacCallum, PharmD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada